CLINICAL TRIAL: NCT01626911
Title: Continuous Regional Arterial Infusion of Low Molecular Weight Heparin in Patients With Severe Acute Pancreatitis
Acronym: CRAI-H
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqin Li, Director of surgical ICU, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAI-H
Record Dates: First submitted 2012-06-16; First posted 2012-06-25 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Acute Pancreatitis
Keywords: severe acute pancreatitis;; continuous regional arterial infusion;; low molecular weight heparin
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRAI (Experimental): CRAI of LMWH in the celiac trunk
  Interventions: Procedure: Continuous regional arterial infusion of low molecular weight heparin in celiac trunk; Other: General treatment
- Conservative treatment (Other): Conservative treatment without CRAI, control group
  Interventions: Other: General treatment

INTERVENTIONS:
Procedure: Continuous regional arterial infusion of low molecular weight heparin in celiac trunk — Put a catheter to the celiac trunk through interventional technique. The approach to celiac trunk was via a femoral artery approach.The tip of the arterial catheter (4F) was placed in celiac trunk which could perfuse the pancreas.After that, continuous infusion of low molecular weight heparin through the catheter will be applied during the first 5 days after placement.
  Arms: CRAI
Other: General treatment — Include fluid resuscitation, percutaneous drainage if needed, antibiotics,organ support, etc.

SUMMARY:
Our animal studies found that continuous regional arterial infusion (CRAI in the celiac trunk) of low molecular weight heparin (LMWH) could alleviate inflammation, improve global hemodynamics and restore organ function in a porcine model of severe acute pancreatitis (SAP,unpublished).

In this study, the investigators aim to evaluate the effects of CRAI of LMWH in the treatment of SAP patients. The investigators suppose CRAI could help improve the outcomes of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of severe acute pancreatitis according to Atlanta criteria
* Within 3 days from the onset of the disease
* Available for interventional treatment(not sensible to radiocontrast agent)

Exclusion Criteria:

* Pregnant pancreatitis
* Receiving surgery or aspiration before;need of early surgery
* Patients with coagulation disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
coagulation related complications | 14 days after the placement of celiac trunk catheter
  bleeding for the most
  coagulative parameters
Pancreatic infection | 28 days

SECONDARY OUTCOMES:
pancreatic necrosis | 28 days
ICU duration | Participants will be followed until the date of discharge from the ICU,assessed up to 6 weeks. Patients who die during hospitalization are excluded from this measurement.
Hospital duration | Participants will be followed until the date of discharge from the hospital,assessed up to 3 months. Patients who die during hospitalization are excluded from this measurement.
Mortality | Participants will be followed until the date of discharge or the date of death from any cause, whichever came first, assessed up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiqin Li, Dr, Principal Investigator — Jinling Hospital, School of Medicine, Nanjing University
Locations (1):
- Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, China, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Lu XS, Qiu F, Li YX, Li JQ, Fan QQ, Zhou RG. Effect of lower-molecular weight heparin in the prevention of pancreatic encephalopathy in the patient with severe acute pancreatitis. Pancreas. 2010 May;39(4):516-9. doi: 10.1097/MPA.0b013e3181c3c954. PMID 20104197